CLINICAL TRIAL: NCT02311348
Title: Comparing Pain in Patients Undergoing Percutaneous Versus Transjugular Techniques of Liver Biopsy
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150025; 15-DK-0025
Record Dates: First submitted 2014-12-05; First posted 2014-12-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2016-12-21

CONDITIONS: Liver Disease
Keywords: Biopsy; Pain
MeSH Terms: conditions — Liver Diseases; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background: In a liver biopsy, a small piece of liver is removed. A percutaneous liver biopsy (PLB) is done through a needle on the right side of your belly. In a transjugular liver biopsy (TLB), the right side of the neck is numbed and a straw-like tube is put in. The tube goes down to your liver and a piece of liver is removed. Researchers want to learn more about the pain people feel after each of these procedures.

Objectives: To compare whether there is more pain associated with the PLB versus TLB.

Eligibility: Adults 18 years or older enrolled in a separate protocol (91-DK-0214) for liver biopsy. They must be able to read, write, and speak English.

Design: Under the separate protocol (91-DK-0214), participants will be screened and have a liver biopsy.

Before the biopsy, participants will give their medical history. They will answer questions about past surgeries and how they feel about pain.

Participants will have a pain test with a device called a dolorimeter. They will sit up with their feet on the ground, and put their thumbs on a table. They will feel pressure on each thumb until it they say it is painful.

Before the biopsy and 2, 4, and 6 hours after the biopsy, they will answer pain questions.

DETAILED DESCRIPTION:
Millions of Americans are diagnosed with some form of Hepatitis or other liver disease requiring treatment. Liver biopsies are frequently performed mainly to stage disease, aid in diagnosis and to guide treatment. As part of the assessment of Hepatitis patients, a liver biopsy is frequently part of the regimen. Liver biopsy procedures can be performed using one of two methods: percutaneous liver biopsy (PLB) or transjugular liver biopsy (TLB). Alknawy & Shiffman (2007) discuss approaches of percutaneous liver biopsy that included the percussion-palpation approach, image guided, ultrasound assisted, ultrasound guided and type of biopsy needle used. The method of liver biopsy selected will not be randomly assigned but will be determined by the hepatologist caring for the patient. Pain can be a complication following a liver biopsy requiring adequate pain management.

Despite an extensive review of previous studies, none were found that discussed the pain experiences of patients who have undergone PLB versus TLB. This study proposes to compare the amount of pain experienced by patients who have undergone PLB versus TLB. Thirty-two male and female patients age 18 years and older who meet study criteria will be invited to participate. The participants will be placed into either the PLB or TLB group with each group consisting of 16 male or 16 female participants. Prior to the biopsy and within the first 6 hours post procedure, at the 2, 4 and 6-hour time points, the patient will be asked to rate their pain on the Visual Analogue Scale (VAS) and on the Numeric Pain Scale (NPS). Additionally, the dolorimeter will be used pre liver biopsy along with the VAS and the NPS as standardized pain measurements.

ELIGIBILITY:
* INCLUSION CRITERIA:

Criteria for subject selection will include the following:

1. 18 years of age or older
2. able to read, write and speak English.
3. capable of providing informed consent
4. subjects undergoing an elective PLB or TLB.
5. baseline pain level will be assessed prior to the liver biopsy using both VAS and NPS.
6. an assessment of pain threshold using a medical device called a dolorimeter.
7. must be enrolled into the 91-DK-0214 protocol

EXCLUSION CRITERIA:

1. patients who are unable to give consent will be excluded from the study.
2. Patient report of a pain level of four or more pre liver biopsy
3. The patient must undergo a baseline pain assessment prior to the liver biopsy using the dolorimeter.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11-20; Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Pain comparison between 2 groups | 0, 2, 4, & 6 hour

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Haynes-Williams, R.N., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States